CLINICAL TRIAL: NCT04627311
Title: Long-term Benefits of Cardiac Rehabilitation Programme
Status: Completed | Type: Observational
Sponsor: Institut d'Assistència Sanitària (Other)
Responsible Party: Sponsor
Other Study IDs: IAssistenciaSanitaria
Record Dates: First submitted 2020-11-08; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Cardiovascular Risk Factor; Cardiac Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A retrospective observational study was conducted on a cohort of 213 patients referred to the Cardiac Rehabilitation programme of Santa "Caterina" Hospital ("Girona", Spain) following acute coronary syndrome (ACS). We evaluated the long-term control of Cardiovascular Risk Factors and the occurrence of major adverse cardiac events (MACE) in a 3-year period of follow-up.

DETAILED DESCRIPTION:
A retrospective observational study was conducted on a cohort of 213 patients referred to the Cardiac Rehabilitation programme of "Santa Caterina" Hospital ("Girona", Spain) following acute coronary syndrome (ACS). We evaluated the long-term control of Cardiovascular Risk Factors and the occurrence of major adverse cardiac events (MACE) in a 3-year period of follow-up.

we found that short-term CVRF control was significantly improved after discharge from the CR unit for all CVRF analysed (LDLc, Systolic blood pressure, tobacco consumption, HbA1C and BMI (body mass index)). Long-term control of low-density lipoprotein cholesterol (LDL-c) and tobacco consumption was maintained from post-CR to year three, although both showed a trend towards deterioration. There was a significant increase in systolic blood pressure and glycosylated haemoglobin (HbA1C) and body mass index (BMI) from post-CR to year three.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in the hospital-based Cardiac Rehabilitation programme of Santa Caterina Hospital of Girona from January 2008, with a 3-year period follow-up.
* Patients diagnosed with ACS - including STEMI, NSTEMI and unstable angina (UA) admitted in the cardiology unit of Santa Caterina Hospital of Girona and Hospital Universitari Dr. Josep Trueta of Girona.
* Patients able to read the information paper and to provide written informed consent of the Cardiac Rehabilitation programme of the Santa Caterina Hospital.

Exclusion Criteria:

* Patients enrolled in the hospital-based Cardiac Rehabilitation programme of Santa Caterina Hospital of Girona with a different diagnosis of heart disease: cardiovascular surgery, congestive heart failure, heart valve disease, etc.
* Data unavailable for a 3-year follow-up study ± 6 months.
* Patients with severe comorbidities or limitation for physical activity, and thus, inability to undergo Cardiac Rehabilitation programmes.
* Stress test with induced significative ischemia with low charge of exercise, arrhythmia induced with the exercise or hypotension response to this.
* Ventricular arrhythmias and other malignant arrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive individuals referred to the hospital-based Cardiac Rehabilitation programme through the Cardiology unit at Santa Caterina Hospital of Girona, after suffering an ACS, with a 3-year period follow-up. A target population of 227 patients were referred to the CR unit during this period. According to inclusion and exclusion criteria, 213 patients were recruited in the retrospective analysis of Girona's health region.
Sampling Method: Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Risk Factors control | 3 years
  To determine whether the control of the CVRF (tobacco consumption, hypertension, hyperlipidaemia, diabetes mellitus type 2 and overweight) is maintained at long term (after 3 years of discharge of the CR unit), among all patients referred to the hospital-based CR programme of Santa "Caterina" Hospital from "Girona" area, after suffering an ACS.

SECONDARY OUTCOMES:
Incidence of Major Adverse Cardiovascular Events (MACE) | 3 years
  To determine the incidence of MACE (Major Adverse Cardiovascular Events:
  ACS, need for revascularization by percutaneous intervention or coronary artery bypass grafting (CABG), stroke, cardiovascular death and/or sudden death) among all patients post-ACS referred to the hospital-based CR programme of Santa "Caterina" Hospital, after 3 years of follow-up.

IPD SHARING:
Plan to Share IPD: No